CLINICAL TRIAL: NCT04847297
Title: Preoperative Biliary Drainage in Malignant Biliary Obstruction - an Observational Cohort Study
Brief Title: Preoperative Biliary Drainage in Malignant Biliary Obstruction
Acronym: PEAR
Status: Not yet recruiting | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Szűcs, Principal Investigator, Associate Professor of the First Surgical Department of the University of Semmelweis, University of Pecs
Other Study IDs: 40393-10/2020/EÜIG
Record Dates: First submitted 2020-12-20; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer
Keywords: pancreatic cancer; biliary drainage; pancreato-duodenectomy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (serum and plasma) from all patients will be stored in the Biobank in order to study laboratory parameters later if required (eg, the laboratory could not measure it), and in order to build up a biobank for later clinical studies to which all participants will be given informed consent. The samples will be stored at -80°C.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative biliary drainage and pancreatoduodenectomy: Patients receiving preoperative biliary drainage before the removal of the tumor.
  Interventions: Procedure: Preoperative drainage and pancreatoduodenectomy
- Pancreatoduodenectomy only: Patients undergoing only surgical intervention, without preoperative drainage.
  Interventions: Procedure: Pancreatoduodenectomy

INTERVENTIONS:
Procedure: Preoperative drainage and pancreatoduodenectomy — Preoperative biliary drainage before surgical removal of the tumor
  Groups: Preoperative biliary drainage and pancreatoduodenectomy
Procedure: Pancreatoduodenectomy — Pancreatic tumor resection without previous preoperative biliary drainage
  Groups: Pancreatoduodenectomy only

SUMMARY:
The first alarming symptom of a malignancy of the pancreas or periampullary tumor can be obstructive jaundice (OJ). Pancreato-duodenectomy (PD) combined with oncological treatment can provide long disease-free survival in resectable cases. The literature regarding the preoperative biliary drainage is controversial. The aim of this multicenter, prospective observational cohort study is to investigate the role of preoperative drainage, and to compare it with surgery alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years
2. OJ of malignant origin (pancreatic head or periampullary tumor)
3. Total bilirubin level ≥ 40 μmol per liter
4. Signed written informed consent

Exclusion Criteria:

1. Proved metastasis
2. Irresectable tumor
3. Neo-adjuvant chemotherapy
4. Co-existing malignancy
5. Pregnancy
6. Patients not fit for resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be patients diagnosed with malignant biliary obstruction who meet all the inclusion criteria but no exclusion criteria. All patients admitted with malignant biliary obstruction with- or without biliary intervention prior to the surgery in the participating hospitals will be assessed for eligibility
Sampling Method: Non-Probability Sample
Enrollment: 353 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of serious complications | 120 days
  rate of serious complications after preoperative biliary drainage and surgery
  1. Pancreatitis
  2. New onset of cholecystitis
  3. Cholangitis
  4. Perforation
  5. Hemorrhage after endoscopic retrograde cholangiopancreatography (ERCP)
  6. Related to stent
     1. Occlusion
     2. Need for exchange Related to surgery
  7. Pancreas anastomosis leakage
rate of serious complications | 120 days
  rate of serious complications after preoperative biliary drainage and surgery defined as:
  1. Pancreatitis
  2. New onset of cholecystitis
  3. Cholangitis
  4. Perforation
  5. Hemorrhage after endoscopic retrograde cholangiopancreatography (ERCP)
  6. Related to stent
     1. Occlusion
     2. Need for exchange Related to surgery
  7. Pancreas anastomosis leakage

SECONDARY OUTCOMES:
Length of hospitalization | 120 days
  Length of hospitalization after biliary drainage and surgery
Mortality | 30 days
  Rate of mortality among groups
Mortality | 120 days
  Rate of mortality among the groups

CONTACTS AND LOCATIONS:
Overall Officials: Péter Hegyi, Study Chair — Insitute for Translational Medicine, University of Pécs, Medical School, Pécs, Hungary; Ákos Szűcs, Principal Investigator — First Surgical Department of the University of Semmelweis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdeldayem H, Ghoneim E, Refaei AA, Abou-Gabal A. Obstructive jaundice promotes intestinal-barrier dysfunction and bacterial translocation: experimental study. Hepatol Int. 2007 Dec;1(4):444-8. doi: 10.1007/s12072-007-9018-1. Epub 2007 Sep 20. PMID 19669340
- [Background] Assimakopoulos SF, Scopa CD, Vagianos CE. Pathophysiology of increased intestinal permeability in obstructive jaundice. World J Gastroenterol. 2007 Dec 28;13(48):6458-64. doi: 10.3748/wjg.v13.i48.6458. PMID 18161914
- [Background] Kuzu MA, Kale IT, Col C, Tekeli A, Tanik A, Koksoy C. Obstructive jaundice promotes bacterial translocation in humans. Hepatogastroenterology. 1999 Jul-Aug;46(28):2159-64. PMID 10521960
- [Background] Ito Y, Bethea NW, Baker GL, McCuskey MK, Urbaschek R, McCuskey RS. Hepatic microcirculatory dysfunction during cholestatic liver injury in rats. Microcirculation. 2003 Oct;10(5):421-32. doi: 10.1038/sj.mn.7800208. PMID 14557825
- [Background] Abraham S, Szabo A, Kaszaki J, Varga R, Eder K, Duda E, Lazar G, Tiszlavicz L, Boros M, Lazar G Jr. Kupffer cell blockade improves the endotoxin-induced microcirculatory inflammatory response in obstructive jaundice. Shock. 2008 Jul;30(1):69-74. doi: 10.1097/SHK.0b013e31815dceea. PMID 18562926
- [Background] Kennedy JA, Clements WD, Kirk SJ, McCaigue MD, Campbell GR, Erwin PJ, Halliday MI, Rowlands BJ. Characterization of the Kupffer cell response to exogenous endotoxin in a rodent model of obstructive jaundice. Br J Surg. 1999 May;86(5):628-33. doi: 10.1046/j.1365-2168.1999.01114.x. PMID 10361183
- [Background] Minter RM, Fan MH, Sun J, Niederbichler A, Ipaktchi K, Arbabi S, Hemmila MR, Remick DG, Wang SC, Su GL. Altered Kupffer cell function in biliary obstruction. Surgery. 2005 Aug;138(2):236-45. doi: 10.1016/j.surg.2005.04.001. PMID 16153432
- [Background] Sheen-Chen SM, Chau P, Harris HW. Obstructive jaundice alters Kupffer cell function independent of bacterial translocation. J Surg Res. 1998 Dec;80(2):205-9. doi: 10.1006/jsre.1998.5467. PMID 9878315
- [Background] Kloek JJ, Heger M, van der Gaag NA, Beuers U, van Gulik TM, Gouma DJ, Levi M. Effect of preoperative biliary drainage on coagulation and fibrinolysis in severe obstructive cholestasis. J Clin Gastroenterol. 2010 Oct;44(9):646-52. doi: 10.1097/MCG.0b013e3181ce5b36. PMID 20142756
- [Background] N Shachiri DK, D Tonev, M Shishenkov. Hemostasiologic Changes during Hepatobiliary Surgery in Patients with Obstructive Jaundice: Pathophysiology and Clinical Considerations. The Internet Journal of Anesthesiology. 2010;28(1).
- [Background] Betjes MG, Bajema I. The pathology of jaundice-related renal insufficiency: cholemic nephrosis revisited. J Nephrol. 2006 Mar-Apr;19(2):229-33. PMID 16736428
- [Background] Uslu A, Tasli FA, Nart A, Postaci H, Aykas A, Bati H, Coskun Y. Human kidney histopathology in acute obstructive jaundice: a prospective study. Eur J Gastroenterol Hepatol. 2010 Dec;22(12):1458-65. doi: 10.1097/MEG.0b013e32833f71f6. PMID 20881503
- [Background] Padillo J, Puente J, Gomez M, Dios F, Naranjo A, Vallejo JA, Mino G, Pera C, Sitges-Serra A. Improved cardiac function in patients with obstructive jaundice after internal biliary drainage: hemodynamic and hormonal assessment. Ann Surg. 2001 Nov;234(5):652-6. doi: 10.1097/00000658-200111000-00010. PMID 11685028
- [Background] Klinkenbijl JH, Jeekel J, Schmitz PI, Rombout PA, Nix GA, Bruining HA, van Blankenstein M. Carcinoma of the pancreas and periampullary region: palliation versus cure. Br J Surg. 1993 Dec;80(12):1575-8. doi: 10.1002/bjs.1800801227. PMID 7507785
- [Background] Trede M, Schwall G. The complications of pancreatectomy. Ann Surg. 1988 Jan;207(1):39-47. doi: 10.1097/00000658-198801000-00009. PMID 3276272
- [Background] Kimmings AN, van Deventer SJ, Obertop H, Rauws EA, Huibregtse K, Gouma DJ. Endotoxin, cytokines, and endotoxin binding proteins in obstructive jaundice and after preoperative biliary drainage. Gut. 2000 May;46(5):725-31. doi: 10.1136/gut.46.5.725. PMID 10764720
- [Background] van der Gaag NA, Kloek JJ, de Castro SM, Busch OR, van Gulik TM, Gouma DJ. Preoperative biliary drainage in patients with obstructive jaundice: history and current status. J Gastrointest Surg. 2009 Apr;13(4):814-20. doi: 10.1007/s11605-008-0618-4. Epub 2008 Aug 23. PMID 18726134
- [Background] Hatfield AR, Tobias R, Terblanche J, Girdwood AH, Fataar S, Harries-Jones R, Kernoff L, Marks IN. Preoperative external biliary drainage in obstructive jaundice. A prospective controlled clinical trial. Lancet. 1982 Oct 23;2(8304):896-9. doi: 10.1016/s0140-6736(82)90866-2. PMID 6126752
- [Background] Pitt HA, Gomes AS, Lois JF, Mann LL, Deutsch LS, Longmire WP Jr. Does preoperative percutaneous biliary drainage reduce operative risk or increase hospital cost? Ann Surg. 1985 May;201(5):545-53. doi: 10.1097/00000658-198505000-00002. PMID 2986562
- [Background] Wig JD, Kumar H, Suri S, Gupta NM. Usefulness of percutaneous transhepatic biliary drainage in patients with surgical jaundice--a prospective randomised study. J Assoc Physicians India. 1999 Mar;47(3):271-4. PMID 10999118
- [Background] Fang Y, Gurusamy KS, Wang Q, Davidson BR, Lin H, Xie X, Wang C. Pre-operative biliary drainage for obstructive jaundice. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD005444. doi: 10.1002/14651858.CD005444.pub3. PMID 22972086
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krle A-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 Statement: defining standard protocol items for clinical trials. Rev Panam Salud Publica. 2015 Dec;38(6):506-14. PMID 27440100
- [Background] Hritz I, Hegyi P. Early Achievable Severity (EASY) index for simple and accurate expedite risk stratification in acute pancreatitis. J Gastrointestin Liver Dis. 2015 Jun;24(2):177-82. doi: 10.15403/jgld.2014.1121.242.easy. PMID 26114177
- [Background] Parniczky A, Mosztbacher D, Zsoldos F, Toth A, Lasztity N, Hegyi P; Hungarian Pancreatic Study Group and the International Association of Pancreatology. Analysis of Pediatric Pancreatitis (APPLE Trial): Pre-Study Protocol of a Multinational Prospective Clinical Trial. Digestion. 2016;93(2):105-10. doi: 10.1159/000441353. Epub 2015 Nov 26. PMID 26613586
- [Background] Zsoldos F, Parniczky A, Mosztbacher D, Toth A, Lasztity N, Hegyi P; Hungarian Pancreatic Study Group and the International Association of Pancreatology. Pain in the Early Phase of Pediatric Pancreatitis (PINEAPPLE Trial): Pre-Study Protocol of a Multinational Prospective Clinical Trial. Digestion. 2016;93(2):121-6. doi: 10.1159/000441352. Epub 2015 Dec 4. PMID 26641250
- [Background] Dubravcsik Z, Madacsy L, Gyokeres T, Vincze A, Szepes Z, Hegyi P, Hritz I, Szepes A; Hungarian Pancreatic Study Group. Preventive pancreatic stents in the management of acute biliary pancreatitis (PREPAST trial): pre-study protocol for a multicenter, prospective, randomized, interventional, controlled trial. Pancreatology. 2015 Mar-Apr;15(2):115-23. doi: 10.1016/j.pan.2015.02.007. Epub 2015 Feb 25. PMID 25754525
- [Background] Marta K, Szabo AN, Pecsi D, Varju P, Bajor J, Godi S, Sarlos P, Miko A, Szemes K, Papp M, Tornai T, Vincze A, Marton Z, Vincze PA, Lanko E, Szentesi A, Molnar T, Hagendorn R, Faluhelyi N, Battyani I, Kelemen D, Papp R, Miseta A, Verzar Z, Lerch MM, Neoptolemos JP, Sahin-Toth M, Petersen OH, Hegyi P; Hungarian Pancreatic Study Group. High versus low energy administration in the early phase of acute pancreatitis (GOULASH trial): protocol of a multicentre randomised double-blind clinical trial. BMJ Open. 2017 Sep 14;7(9):e015874. doi: 10.1136/bmjopen-2017-015874. PMID 28912191
- [Background] Dubravcsik Z, Farkas G, Hegyi P, Hritz I, Kelemen D, Lasztity N, Morvay Z, Olah A, Pap A, Parniczky A, Sahin-Toth M, Szentkereszti Z, Szmola R, Takacs T, Tiszlavicz L, Szucs A, Czako L; Magyar Hasnyalmirigy Munkacsoport, Hungarian Pancreatic Study Group. [Autoimmune pancreatitis. Evidence based management guidelines of the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 22;156(8):292-307. doi: 10.1556/OH.2015.30061. Hungarian. PMID 25662147
- [Background] Hritz I, Czako L, Dubravcsik Z, Farkas G, Kelemen D, Lasztity N, Morvay Z, Olah A, Pap A, Parniczky A, Sahin-Toth M, Szentkereszti Z, Szmola R, Szucs A, Takacs T, Tiszlavicz L, Hegyi P; Magyar Hasnyalmirigy Munkacsoport, Hungarian Pancreatic Study Group. [Acute pancreatitis. Evidence-based practice guidelines, prepared by the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 15;156(7):244-61. doi: 10.1556/OH.2015.30059. Hungarian. PMID 25661970
- [Background] Szmola R, Farkas G, Hegyi P, Czako L, Dubravcsik Z, Hritz I, Kelemen D, Lasztity N, Morvay Z, Olah A, Parniczky A, Rubovszky G, Sahin-Toth M, Szentkereszti Z, Szucs A, Takacs T, Tiszlavicz L, Pap A; Magyar Hasnyalmirigy Munkacsoport, Hungarian Pancreatic Study Group. [Pancreatic cancer. Evidence based management guidelines of the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 22;156(8):326-39. doi: 10.1556/OH.2015.30063. Hungarian. PMID 25662149
- [Background] Takacs T, Czako L, Dubravcsik Z, Farkas G, Hegyi P, Hritz I, Kelemen D, Lasztity N, Morvay Z, Olah A, Pap A, Parniczky A, Patai A, Sahin-Toth M, Szentkereszti Z, Szmola R, Tiszlavicz L, Szucs A; Magyar Hasnyalmirigy Munkacsoport. [Chronic pancreatitis. Evidence based management guidelines of the Hungarian Pancreatic Study Group]. Orv Hetil. 2015 Feb 15;156(7):262-88. doi: 10.1556/OH.2015.30060. Hungarian. PMID 25661971
- [Background] van der Gaag NA, Rauws EA, van Eijck CH, Bruno MJ, van der Harst E, Kubben FJ, Gerritsen JJ, Greve JW, Gerhards MF, de Hingh IH, Klinkenbijl JH, Nio CY, de Castro SM, Busch OR, van Gulik TM, Bossuyt PM, Gouma DJ. Preoperative biliary drainage for cancer of the head of the pancreas. N Engl J Med. 2010 Jan 14;362(2):129-37. doi: 10.1056/NEJMoa0903230. PMID 20071702
- [Background] Sewnath ME, Karsten TM, Prins MH, Rauws EJ, Obertop H, Gouma DJ. A meta-analysis on the efficacy of preoperative biliary drainage for tumors causing obstructive jaundice. Ann Surg. 2002 Jul;236(1):17-27. doi: 10.1097/00000658-200207000-00005. PMID 12131081
- [Background] Sun C, Yan G, Li Z, Tzeng CM. A meta-analysis of the effect of preoperative biliary stenting on patients with obstructive jaundice. Medicine (Baltimore). 2014 Nov;93(26):e189. doi: 10.1097/MD.0000000000000189. PMID 25474436